CLINICAL TRIAL: NCT01594632
Title: A Study to Evaluate the Contraceptive Effectiveness, Safety and Acceptability of Sino-implant II
Brief Title: Safety,Effectiveness and Acceptability of Sino-implant II in DR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10242
Record Dates: First submitted 2011-10-13; First posted 2012-05-09 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Contraception
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonization; IND Investigational New Drug Application; IRB Institutional Review Board; IU International units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jadelle (Experimental): Contraception using Jadelle implant
  Interventions: Drug: Jadelle
- Sino-implant (II) (Active Comparator): levonorgestrel containing subdermal contraceptive implant [Zarin, Femplant, Trust or Simplant]
  Interventions: Drug: Sino-implant (II)

INTERVENTIONS:
Drug: Jadelle — LNG containing subdermal contraceptive implant
  Arms: Jadelle
Drug: Sino-implant (II) — LNG containing subdermal contraceptive implant
  Other Names: Zarin, Femplant, Trust, Simplant
  Arms: Sino-implant (II)

SUMMARY:
A study to assess the contraceptive effectiveness of Sino-implant (II).

DETAILED DESCRIPTION:
Randomized trial to assess the contraceptive effectiveness of Sino-implant (II) and to compare levonorgestrel concentrations, safety and acceptability of Sino-implant (II) and Jadelle.

ELIGIBILITY:
Inclusion Criteria:• In good general health

* Aged between 18 and 44 years, inclusive
* Not pregnant
* Not lactating
* Not wishing to become pregnant in the next five years
* Request long-acting reversible contraception
* If previously used injectable contraceptives for pregnancy prevention, be more than 9 months since last injection of Depo-Provera and more than 3 months after the last injection of a combined injectable contraceptive
* If previously used LNG-containing oral pills or implants, be more than 1 week after last hormone intake or implant removal
* Be able to understand the information provided and to make personal decisions on participation
* Consent to participation and sign a consent form
* Agree and be able to return to the clinic for follow-up visits over five years

Exclusion Criteria:

* acute deep venous thrombosis and/or pulmonary embolism or history of thromboembolic disease
* systemic lupus erythematosus with positive or unknown antiphospholipid antibodies
* unexplained vaginal bleeding
* current or history of breast cancer
* acute liver disease or cirrhosis
* benign or malignant tumor of the liver
* use of rifampicin, and/or anticonvulsants (barbiturates, phenytoin, phenobarbital, carbamazepine, oxcarbazepine, primidone, topiramate), and/or herbal products containing St. John's Wort (Hypericum perforatum)
* more than one sexual partner in the last 3 months
* diagnosis or treatment for a sexually transmitted infection (STI) within the past 30 days for her or partner (excluding recurrent genital herpes or condyloma)
* known HIV positive status for her or partner
* any condition (social or medical) which in the opinion of the Investigator would make study participation unsafe, would interfere with adherence to study requirements or complicate data interpretation
* BMI greater than or equal to 30 (for the sub-group of women with intensive LNG sampling)

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 650 (Actual)
Dates: Start 2011-01; Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the contraceptive effectiveness of Sino-implant (II) during 4 years of use. | 4 years
  Pearl Index (number of pregnancies per 100 woman-years) over 4 years of use of Sino-implant (II).

SECONDARY OUTCOMES:
Evaluate the contraceptive effectiveness of Sino-implant (II) during 5 years of use | 5 years
  Pearl Index over 5 years of use of Sino-implant (II) ; continuation & reasons for discontinuation in both groups.
Compare concentrations of levonorgestrel through 5 years after insertion of Sino-implant (II) and Jadelle | 5 years
  annual and cumulative probability of pregnancy during 5 years of use of Sino-implant (II);
Compare pharmacokinetic profiles of Sino-implant (II) and Jadelle during the first 6 months of use in a sub-group of users undergoing intensive levonorgestrel sampling | 5 years
  The PK profile of LNG during the first 6 months post-insertion including the following parameters in a sub-group of users undergoing intensive LNG sampling:
  Mean LNG concentrations at 6 hours, 24 hours, 48 hours, 72 hours, 7 days and 90 days post-insertion Concentration-time profiles of LNG (individual and pooled) Maximal concentration (Cmax) and time to maximal concentration (Tmax) AUC0-7 days, AUC0-1mon, AUC0-3mon and AUC0-6mon
Compare the safety and acceptability of Sino-implant (II) and Jadelle during 5 years of use | 5 years
  Adverse event rates in both treatment groups Annual and cumulative probability of early discontinuation in both treatment groups Reasons for discontinuation in both treatment groups Responses on acceptability questionnaires in both treatment groups
Compare free levonorgestrel index through 5 years after insertion of Sino-implant (II) and Jadelle in a sub-group of approximately 150 users. | 5 years
  free levonorgestrel index, estimated as the ratio of levonorgestrel to sex hormone binding globulin at various point during 5 years of product use in a sub-group of approximately 150 women.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Brache, LIC, Principal Investigator — Profamilia
Locations (1):
- Profamilia, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Undecided